CLINICAL TRIAL: NCT06597786
Title: Neoadjuvant Exercise Therapy in Solid Tumors: A Phase 1b Dose Expansion Trial
Brief Title: A Study of Exercise Therapy in People With Solid Tumor Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Focusing on other studies
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-232
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Solid Tumor Cancer
Keywords: Exercise Therapy; 24-232
MeSH Terms: interventions — Exercise Therapy

STUDY DESIGN:
Intervention Model Description: A single-center, open-label, phase 1b dose-expansion trial of neoadjuvant (preoperative) exercise therapy in patients with prespecified solid tumors.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise therapy (Experimental): Exercise therapy will comprise individualized treadmill walking delivered up to 5 times weekly (over a 7-day period) to achieve a weekly cumulative dose of 225 minutes per week. The minimum treatment period will be 3 weeks. Exercise therapy will be administered via a patient-centric, decentralized platform: Digital Platform for Exercise (DPEx). DPEx will permit all study procedures to be conducted remotely in patients' homes.
  Interventions: Other: Exercise therapy

INTERVENTIONS:
Other: Exercise therapy — Patients will receive a study kit which includes a smart watch (for monitoring of mobility / lifestyle patterns), heart rate monitor, blood pressure cuff, scale, and e-tablet. Patients may receive a treadmill to perform exercise therapy sessions. The treadmills and study kits are MSK owned equipment that will be deployed to the patients' homes and returned at the end of the study.

SUMMARY:
The purpose of this study is to find out whether exercise therapy is an effective and safe treatment that causes few or mild side effects when done before standard surgery for solid tumor cancer. The researchers will also study whether the program is feasible (practical) by tracking how well participants follow the program.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed (on preoperative biopsy), resectable, treatment naïve cancer of one of the following types: head and neck, lung, renal, liver, colorectal, gastric, ovarian, melanoma, pancreas, or breast cancer.
* Age ≥18 years.
* An interval of ≥3 weeks until planned surgical resection; surgery will not be delayed to accommodate the minimum length of exercise therapy intervention in any circumstance.
* Measurable disease based on standard of care radiology scans or confirmation by the surgeon.
* Body weight ≤ 385 lbs (≤ 174 kg)
* Non-exercisers, defined as ≤60 minutes of moderate or vigorous exercise/week based on self-report using a validated survey.
* Cleared for moderate-intensity exercise therapy using the Physical Activity Readiness Questionnaire (PAR-Q)+ with screening clearance provided at the discretion of the PI/exercise physiologist.
* Willingness to comply with all study-related procedures

Exclusion Criteria:

* Distant metastases.
* Receiving any form of antitumor therapy.
* Enrollment onto any other interventional investigational study except interventions determined by the PI not to confound the effect of exercise on study outcomes.
* Any other diagnosis of invasive cancer currently requiring active treatment.
* Any other condition (e.g., pregnancy) or intercurrent illness that, in the opinion of the investigator, makes the subject a poor candidate for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-09-12 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
change in Ki67 values | up to 3 years
  With at least one pretreatment (baseline) or postintervention measurement of Ki67 will be considered evaluable. To characterize biological activity of neoadjuvant exercise therapy as defined by the change in tumor cell proliferation marker (Ki67) evaluated in paired formalin-fixed paraffin embedded (FFPE) tumor samples obtained before (diagnostic biopsy) and after (surgical resection) exercise therapy. The biopsies will be collected as part of the standard medical care.

CONTACTS AND LOCATIONS:
Overall Officials: Lee Jones, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm